CLINICAL TRIAL: NCT03126513
Title: Safety and Efficacy of Gastric Per Oral Endoscopic Myotomy (G-POEM) in Patients With Refractory Gastroparesis
Brief Title: Gastric Per Oral Endoscopic Myotomy (G-POEM) in Refractory Gastroparesis
Acronym: G-POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2017-3601-45
Record Dates: First submitted 2017-04-18; First posted 2017-04-24 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Gastroparesis Postoperative; Gastroparesis Due to Diabetes Mellitus; Idiopathic Gastric Stasis
Keywords: G-POEM; Safety; Efficacy
MeSH Terms: interventions — Pyloromyotomy

STUDY DESIGN:
Intervention Model Description: This a prospective study that evaluates G-POEM in a group of participants with diagnosis of refractory gastroparesis. Participants are sequentially recruited as diagnosed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- G-POEM in refractory gastroparesis (Experimental): Participants with refractory gastroparesis will be confirmed by endoscopy, clinical and scintigraphy studies.
  Interventions: Procedure: G-POEM

INTERVENTIONS:
Procedure: G-POEM — After confirmation of refractory gastroparesis, participants will undergo to gastric POEM. Participants will be admitted to hospital 24hrs before procedure and IV antibiotics will be given and then the procedure will be done. Technique consist of 4 steps: First: a submucosa injection of saline solution with methylene blue at 3-4cms from pylorus. Second: a submucosa incision and tunnel creation up to pyloric area. Third: Myotomy of the circular and longitudinal muscular layers of the pylorus and the antrum. Fourth: closure of the mucosal incision with hemoclips. After procedure they will be kept on surveillance and will be followed-up with clinical, endoscopic and scintigraphic studies up to 1 year after procedure.
  Other Names: Gastric per-oral endoscopic myotomy

SUMMARY:
Refractory gastroparesis is a disease characterized by a delayed gastric emptying without a mechanical obstruction. Actual treatments have a limited efficacy and gastric per-oral endoscopic myotomy (G-POEM) is a new treatment that has demonstrated initial promising results in these patients. The investigators aims are to evaluate security and efficacy of this endoscopic treatment in participants with refractory gastroparesis.

DETAILED DESCRIPTION:
Gastroparesis is a chronic, condition characterized by a delayed gastric emptying without a mechanical obstruction. This disease is associated with high morbidity and mortality with a prevalence up to 4% of population. Patients with this disease have a reduced quality of life. The principal etiologies include: post-surgical, diabetes, medications and idiopathic. Symptoms include nausea, vomiting, early satiety, bloating and abdominal pain. Diagnosis is based on the combination of symptoms and studies as gastroscopy that shows retained food in the stomach without a gastric outlet obstruction and confirmed with a gastric emptying scintigraphy. Treatments have limited effect in these patients, including medications, botulinum toxin injection, surgical gastric electrical stimulation, laparoscopic pyloroplasty and stent placement. G-POEM is a new technique based on per-oral endoscopic myotomy treatment in achalasia patients, which has been recently proposed for treatment of patients with refractory gastroparesis with good initial results. The investigators aim is to evaluate the safety and efficacy of this new technique in a group of mexican participants with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory gastroparesis based on delayed gastric emptying symptoms: Nausea, retching, vomiting, abdominal pain, early satiety, post-prandial fullness, bloating.
* Refractoriness defines as the presence of symptoms with failure or recurrence after other type of treatment.
* Any etiology: diabetes, post-surgical, idiopathic

Exclusion Criteria:

* Pregnancy
* Portal hypertension
* Gastric malignant condition
* Active prepyloric ulcer
* Mechanical pyloric stenosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Efficacy of G-POEM in gastroparesis in percentage of scintigraphic improvement at 4hrs | 1, 6 and 12 months
  The investigators will compare the percentage of improvement in scintigraphy before and after procedure

SECONDARY OUTCOMES:
security of G-POEM in gastroparesis | up to 30 days after procedure
  measured as the presence of complications during or after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernandez, MD, Principal Investigator — IMSS
Locations (1):
- Centro Medico Nacional Siglo XXI Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahuja NK, Clarke JO. Pyloric Therapies for Gastroparesis. Curr Treat Options Gastroenterol. 2017 Mar;15(1):230-240. doi: 10.1007/s11938-017-0124-4. PMID 28124202
- [Result] Khashab MA, Ngamruengphong S, Carr-Locke D, Bapaye A, Benias PC, Serouya S, Dorwat S, Chaves DM, Artifon E, de Moura EG, Kumbhari V, Chavez YH, Bukhari M, Hajiyeva G, Ismail A, Chen YI, Chung H. Gastric per-oral endoscopic myotomy for refractory gastroparesis: results from the first multicenter study on endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2017 Jan;85(1):123-128. doi: 10.1016/j.gie.2016.06.048. Epub 2016 Jun 25. PMID 27354102
- [Result] Mekaroonkamol P, Li LY, Dacha S, Xu Y, Keilin SD, Willingham FF, Cai Q. Gastric peroral endoscopic pyloromyotomy (G-POEM) as a salvage therapy for refractory gastroparesis: a case series of different subtypes. Neurogastroenterol Motil. 2016 Aug;28(8):1272-7. doi: 10.1111/nmo.12854. Epub 2016 May 15. PMID 27197717
- [Result] Xue HB, Fan HZ, Meng XM, Cristofaro S, Mekaroonkamol P, Dacha S, Li LY, Fu XL, Zhan SH, Cai Q. Fluoroscopy-guided gastric peroral endoscopic pyloromyotomy (G-POEM): a more reliable and efficient method for treatment of refractory gastroparesis. Surg Endosc. 2017 Nov;31(11):4617-4624. doi: 10.1007/s00464-017-5524-y. Epub 2017 Apr 13. PMID 28409375
- [Result] Geyl S, Legros R, Charissou A, Mesturoux L, Couquet CY, Carrier P, Brayette A, El-Ouafi Z, Loustaud-Ratti V, Sautereau D, Monteil J, Jacques J. Peroral endoscopic pyloromyotomy accelerates gastric emptying in healthy pigs: proof of concept. Endosc Int Open. 2016 Jul;4(7):E796-9. doi: 10.1055/s-0042-108192. Epub 2016 Jun 29. PMID 27556100
- [Result] Gonzalez JM, Lestelle V, Benezech A, Cohen J, Vitton V, Grimaud JC, Barthet M. Gastric per-oral endoscopic myotomy with antropyloromyotomy in the treatment of refractory gastroparesis: clinical experience with follow-up and scintigraphic evaluation (with video). Gastrointest Endosc. 2017 Jan;85(1):132-139. doi: 10.1016/j.gie.2016.07.050. Epub 2016 Jul 28. PMID 27478028